CLINICAL TRIAL: NCT01437527
Title: Body Image Therapy in Anorexia Nervosa
Acronym: PIPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D465; 2010-A01427-32 (Other: Afssaps)
Record Dates: First submitted 2011-09-20; First posted 2011-09-21 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; CMME-TCA Unit; Centre Hospitalier Sainte Anne
MeSH Terms: conditions — Anorexia Nervosa | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional arm (Experimental): Body image therapy with Anamorphic Micro software
  Interventions: Behavioral: Anamorphic Micro software
- control arm (Active Comparator): Body image therapy as usual
  Interventions: Behavioral: therapy as usual

INTERVENTIONS:
Behavioral: Anamorphic Micro software — Body image therapy with Anamorphic Micro software
  Arms: Interventional arm
Behavioral: therapy as usual — Body image therapy as usual
  Arms: control arm

SUMMARY:
The purpose of the study is to test a new procedure of body image therapy in anorexia nervosa, using the anamorphic micro software.

DETAILED DESCRIPTION:
Anorexia nervosa is a severe psychiatric disorder, with high level of mortality and hospitalization is often necessary for the treatment of severe and/or chronic cases.

Anorexic patients often experience a serious disturbance in body and their own shape perception. Body image work should be enhanced in the treatment of anorexia nervosa.

The aim of the study is to test a new body image therapy using the anamorphic Micro software.

Ten sessions of assessment of the patient's own shape and of correction of distorted perceptions of body size with Anamorphic Micro software will be compared to ten sessions of body image therapy as usual.

French 100 anorexia women hospitalized in a specialized Eating Disorder Unit will participate to the study, randomized in 2 arms :

* Body image therapy with Anamorphic Micro software
* Body image therapy as usual

ELIGIBILITY:
Inclusion Criteria:

* woman
* more than 18 years old
* anorexia nervosa
* hospitalized in the CMME (CHSA) TCA Unit
* Body Mass Index ≥ 16
* Informed consent

Exclusion Criteria:

* pregnancy
* severe motor, sensitive or sensorial impairment
* no affiliation of national health service
* dependent of a trusteeship or guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Body Shape Questionnaire | after the 10 sessions of body image therapy
  Body Shape Questionnaire Score after the 10 sessions of body image therapy

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra PHAM - SCOTTEZ, MD, Principal Investigator — Centre Hospitalier Sainte Anne
Locations (1):
- Centre Hospitalier Sainte Anne, Paris, France